CLINICAL TRIAL: NCT04067687
Title: Palliative Intervention to Improve Quality of Life in Children With Cancer: A Randomized Controlled Trial
Brief Title: Home Visit Intervention in Pediatric Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Murti Andriastuti, Doctor, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PedPalliative01
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Pediatric Cancer; Palliative
Keywords: palliative; cancer; pediatric
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Two arm of control group and intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No palliative home visit intervention
- Intervention (Experimental): Palliative home visit intervention
  Interventions: Other: Palliative home visit

INTERVENTIONS:
Other: Palliative home visit — a 3-month home visit, providing two-way communication between a trained health worker and patients with or without their parents were conducted as the intervention (report by proxy or self-report). Interventions were given in 6 sessions (1 session every 2 weeks) focusing on problems solving education, symptoms management, self-care, communication, decision making, and long-term care plan assistance.
  Arms: Intervention

SUMMARY:
A randomized controlled trial to compare the quality of life between participants who were given palliative care (a 3-month home visit) and those who were not (intervention vs control group) was conducted. Participants consisted of children with cancer aged 2-18 years old. A two-way communication between a trained health worker and participants with or without their parents were conducted as the intervention (report by proxy or self-report). Interventions were given in 6 sessions (1 session every 2 weeks) focusing on problems solving education, symptoms management, self-care, communication, decision making, and long-term care plan assistance. In the first and twelfth week of the intervention, all participants were assessed with the Pediatric Quality of Life Inventory (PedsQLTM) questionnaire cancer module 3.0. Symptomps intensityof anorexia, sleep diturbance, and pain will be asessed in each visit. Participants were followed, Emergency Room (ER) admissions were recorded during follow up period. During the follow up period, ER admissions were recorded further.

ELIGIBILITY:
Inclusion Criteria:

* Child age 2-18 years old with malignancies who undergo treatments at the Department of Child Health of Cipto Mangunkusumo Hospital, during the study period.
* All participants who meet the criteria to get palliative care, participants with a total score ≥ 4 based on palliative screening form.
* Participants and or parents agree to be enrolled in study

Exclusion Criteria:

* Patients who live outside Jakarta and therefore unreachable to get palliative intervention

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of life cancer child | at the end of 3 months follow up
  Measured using PedsQLTM cancer module 3.0 that consisted of eight dimension. Each dimension consisted of several items to be answered. Item scaling was answered in 5-point Likert scale from 0 (Never) to 4 (Almost always). Scores are transformed to a 0 to 100 scale. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. If more than 50% of the items in the scale are missing, the scale scores should not be computed. Mean score = Sum of the items over the number of items answered. Total score is acquired by summing of all the items over the number of items answered on all the Scales.Higher scores indicate lower problems.

SECONDARY OUTCOMES:
Emergency room visits | during 3 months follow up
  Frequency of emergency room visit is recorded during 3-months follow up period. Total number of emergency rom visits will be summed.
Symptomps intensity | during 3 months follow up
  Measured using Edmonton Symptoms Asessment Scale. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity. The patient and family should be taught how to complete the scales. Mean score is acquired by summing all scores then divided it by total number of assesment.

CONTACTS AND LOCATIONS:
Overall Officials: Murti Andriastuti, Doctor, Principal Investigator — Indonesia University, Cipto Mangunkusumo Hospital Jakarta
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No